CLINICAL TRIAL: NCT06924684
Title: Efficacy Of High-Dose Rosuvastatin Preloading Before Primary Percutaneous Coronary Intervention In Patients Suffering From St-Elevation Myocardial Infarction
Brief Title: High-Dose Rosuvastatin Preloading for Enhanced Outcomes in STEMI Patients Undergoing Primary PCI
Acronym: HEROS-PCI
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheikh Zayed Federal Postgraduate Medical Institute (Other)
Collaborators: Punjab Institute of Cardology (Other)
Responsible Party: Principal Investigator, Sohaib Ashraf, Senior Registrar, Deparment of Cardiology, Principal Investigator, Sheikh Zayed Federal Postgraduate Medical Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UHS/IRB/0156/2024
Record Dates: First submitted 2024-12-30; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-12

CONDITIONS: ST Elevation (STEMI) Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Active Comparator): Tab Rosuvastatin 40mg at presentation. Tab Rosuvastatin 20mg at night for 30 days.
  Interventions: Drug: Statin monotherapy (rosuvastatin or atorvastatin)
- Placebo Arm (Placebo Comparator): Placebo capsule 40mg (weight) at presentation. Tab Rosuvastatin 20mg at night for 30 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Statin monotherapy (rosuvastatin or atorvastatin) — Tab Rosuvastatin 40mg (weight) at presentation. Tab Rosuvastatin 20mg at night for 30 days.
  Other Names: Rosuvastatins
  Arms: Intervention arm
Drug: Placebo — Placebo caspule
  Arms: Placebo Arm

SUMMARY:
To compare the efficacy of high dose rosuvastatin preloading vs placebo before primary PCI in terms of MACE at 30 days

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years Patients undergoing primary angiography

Exclusion Criteria:

* Hemodynamically unstable patients. History or clinical evidence of any co-morbidities. Taking any medications regularly even statins.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-06-23 (Estimated); Study Completion 2025-07-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of MACE | 30 days
In-Hospital mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Sohaib Ashraf, MD, Principal Investigator — Shaikh Zayed Hospital
Locations (2):
- Pakistan (2):
  - Shaikh Zayed Hsopital, Lahore
  - Punjab Institute of Cardiology, Lahore